CLINICAL TRIAL: NCT02717962
Title: Phase 2 Study of VAL-083 Treatment for MGMT Unmethylated Bevacizumab-naïve Glioblastoma in the Adjuvant or Recurrent Setting
Brief Title: Study of VAL-083 in Patients With MGMT Unmethylated, Bevacizumab-naive Glioblastoma in the Adjuvant or Recurrent Setting
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Kintara Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DLM-16-001
Expanded Access: NCT03138629 (No longer available)
Record Dates: First submitted 2016-03-16; First posted 2016-03-24 (Estimated); Last update posted 2025-08-29 (Actual); Status verified 2025-08

CONDITIONS: Glioma; Glioblastoma; Glioblastoma Multiforme; GBM; Brain Cancer
Keywords: Glioma; Glioblastoma; Glioblastoma multiforme; GBM; brain tumor; brain cancer; recurrent brain tumor; recurrent brain cancer; refractory brain tumor; refractory brain cancer; recurrent GBM; refractory GBM; recurrent glioma; refractory glioma; recurrent glioblastoma; refractory glioblastoma; recurrent glioblastoma multiforme; refractory glioblastoma multiforme; failed bevacizumab; temodar failure; temozolomide failure; adjuvant therapy
MeSH Terms: conditions — Glioma; Glioblastoma; Brain Neoplasms | interventions — Dianhydrogalactitol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- VAL-083, Dianhydrogalactitol (Group 1) (Experimental): Patients with recurrent/progressive GBM
  Interventions: Drug: VAL-083, Dianhydrogalactitol
- VAL-083, Dianhydrogalactitol (Group 2) (Experimental): Newly diagnosed GBM patients who have completed chemoradiation treatment with temozolomide and received no subsequent maintenance temozolomide
  Interventions: Drug: VAL-083, Dianhydrogalactitol

INTERVENTIONS:
Drug: VAL-083, Dianhydrogalactitol — The dosing regimen for patients will be VAL-083 (30 mg/m2) administered IV for 3 consecutive days at the beginning of every 21-day cycle. Patients will continue to receive VAL 083, for up to 12, 21-day treatment cycles or until they fulfill one of the criteria for study discontinuation.

SUMMARY:
The purpose of this phase 2, two arm, biomarker-driven study is to determine if treatment of O-6-methylguanine-DNA methyltransferase (MGMT) unmethylated glioblastoma with VAL-083 improves overall survival (OS), compared to historical control, in the adjuvant or recurrent setting.

DETAILED DESCRIPTION:
Recurrent GBM is characterized by a dismal prognosis, with a median overall survival of 6.9 months. While a standard of care is established for the initial treatment of GBM - radiation with concurrent and adjuvant temozolomide chemotherapy - management of recurrent disease (NCCN, 2014) remains suboptimal. Treatment options include repeat surgery, re-irradiation, or chemotherapy (including experimental targeted therapies, biologic agents, and immunotherapies). Only a minority of patients has response to these treatments, and the resultant benefits in progression-free and overall survival are in the order of weeks to months.

Prognosis and response to therapy are known to be better in patients with a methylated MGMT promoter gene. Epigenetic silencing of MGMT by promoter methylation is an important factor in predicting outcome for patients with GBM treated with temozolomide. Approximately 66% of GBM tumors are MGMT unmethylated (high expression of MGMT), which through a MGMT repair mechanism, confers resistance to temozolomide, the standard chemotherapy treatment of GBM.

VAL-083, Dianhydrogalactitol (DAG), unlike temozolomide, is demonstrated to be active independent of MGMT resistance mechanisms, in vitro. Thus, it may provide a treatment option for those patients that are considered likely to be poor responders to temozolomide.

This is a non-comparative, two arm, biomarker-driven study with VAL-083 in GBM patients with either recurrent disease (Group 1) or newly diagnosed GBM patients requiring maintenance therapy after chemoradiation with temozolomide (Group 2).

Group 1: A total of up to 83 patients with recurrent/progressive GBM will be enrolled. This will include 35 patients treated at 40 mg/m2 and up to 48 patients treated at 30 mg/m2.

Group 2: Up to an additional 36 newly diagnosed GBM patients who have completed chemoradiation treatment with temozolomide and received no subsequent maintenance temozolomide will be enrolled.

Eligible patients will receive VAL-083 IV on days 1, 2, and 3, for up to 12, 21-day treatment cycles or until they fulfill one of the criteria for study discontinuation (disease progression, death, intolerable toxicities, investigator's judgment, or withdrawal of consent). Disease status will be evaluated with clinical and MRI evaluation every other 21-day cycle, while the patient is receiving VAL-083 treatment, and then approximately every 42 ± 7 days while remaining on study. Symptom burden will be evaluated using the MD Anderson Symptom Inventory-Brain Tumor (MDASI-BT) completed by patients at baseline and at the time of each imaging evaluation.

Interval medical histories, targeted physical exams, neurologic evaluations, complete blood counts, and other laboratory and safety assessments will be performed approximately every 21-days. Blood samples will be taken at Cycle 1 Day 1 pre-dose, 15 ± 5 min, 30 ± 5 min, 60 ± 10 min, 120 ± 10 min, 240 ± 15 min, and 360 ± 15 min after the end of the of iv infusion with VAL-083 to determine the PK profile and dose-exposure relationship of VAL-083.

Toxicity will be evaluated and documented using the NCI CTCAE version 4.

This study will take approximately 36 months to enroll.

ELIGIBILITY:
General Inclusion Criteria:

* Patient must willingly provide written consent after being informed of the procedure to be followed, the experimental nature of the therapy, alternatives, potential benefits, side effects, risks, and discomforts.
* Patients must be ≥ 18 years old.
* Patients must have histologically confirmed initial diagnosis of primary intracranial WHO Grade IV malignant glioma (glioblastoma).
* Patients must have preliminary GBM MGMT status (tumor must be MGMT promoter unmethylated) determined prior to study entry. If initial MGMT status is determined to be "unmethylated", by an outside institution the patient may be enrolled and begin treatment. However, MGMT status must be retested following enrollment by central laboratory CLIA certified testing at MD Anderson.
* Patients must have Karnofsky Performance Status (KPS) > 60% (i.e., 70, 80, 90 or 100).
* Adequate recovery from all recent surgery is required. At least 21-days must have elapsed from the time of any major surgery, including craniotomy/tumor resection. Patients must have recovered from all surgery-related toxicities to Grade 1 or less.
* Prior therapy with gamma knife or other focal high-dose radiation is allowed, but at least 2 weeks must have elapsed from the time of treatment, and the patient must have subsequent histologic documentation of recurrence, unless the recurrence is a new lesion outside the irradiated field.
* Patients having prior therapy with Laser Induced Thermal Therapy (LITT) is allowed, but at least 21 days must have elapsed from last LITT, with recovery from all LITT-related toxicities to Grade 1 or less and subsequent histologic documentation of recurrence
* Patients must be at least 4 weeks from last dose of chemotherapy.
* Patients must have recovered from all treatment-related toxicities to Grade 1 or less.
* If receiving corticosteroids, patients must be on a stable or decreasing dose of corticosteroids for ≥ 5 days prior to baseline MRI.
* Patients must have a predicted life expectancy of at least 12 weeks.
* Patients must have adequate bone marrow and organ function.
* Patients must be willing and able to comply with scheduled visits, treatment plan, and laboratory tests and accessible for follow-up after treatment termination.
* If the patient has been using the Optune™ device, it will be discontinued before initiating treatment with either study medication, and per inclusion criterion listed above, the patient must have recovered from all treatment-related toxicities to Grade 1 or less.
* Pregnancy restrictions - Women of childbearing potential must have a negative B-HCG documented within 7 days prior to registration

Group Specific Inclusion Criteria - Recurrent GBM (Group 1):

* Patients must have recurrent disease whose initial diagnostic pathology confirmed glioblastoma will not need re-biopsy. Alternately, patients with prior intracranial low-grade glioma or anaplastic glioma will be eligible, if histologic assessment demonstrates transformation to GBM (first diagnosis of secondary GBM).
* Patients must have radiographic evidence of recurrent/progressive GBM after prior therapy (biopsy or resection and chemoradiation); 1st recurrence of GBM only, per RANO criteria. Histologically documented transformation from a lower grade gliomas will be considered first recurrence.
* Patients must be >12 weeks from radiotherapy, to minimize the potential for MRI changes related to treatment (pseudoprogression) that might be misdiagnosed as true progression of disease, unless the patient fulfills criteria for early progressive disease by RANO.
* Patients must have been previously treated for GBM with concurrent temozolomide and radiation followed by adjuvant temozolomide chemotherapy.
* Patients must be at least 4 weeks or 5 half-lives (whichever is shorter) from the last dose of prior investigational anti-cancer drugs.

Group Specific Inclusion Criteria - Newly Diagnosed GBM requiring maintenance therapy (Group 2)

* Patients must not have recurrent disease.
* Patients must be < 6 weeks from radiotherapy to start of treatment with VAL-083.
* Patients must have been previously treated for GBM with concurrent temozolomide and radiation, and received no subsequent maintenance temozolomide chemotherapy.
* No prior investigational agent.

Exclusion Criteria:

* Within 12 weeks of chemoradiation unless the patient fulfills criteria for early progressive disease by RANO, for Group 1; and, more than 6 weeks from chemoradiation for Group 2.
* Receipt of investigational agents within 5 half-lives of last dose of investigational agent.
* Concurrent use of other investigational agents or Optune™ device
* Prior therapy with lomustine.
* Prior therapy with bevacizumab.
* Current history of neoplasm other than the entry diagnosis. Patients with previous cancers treated and cured with local therapy alone may be considered with approval of the Sponsor.
* Evidence of leptomeningeal spread of disease.
* Need for urgent palliative intervention (e.g., impending herniation).
* Severe, intercurrent illness including, but not limited to unstable systemic disease, including ongoing or active infection, uncontrolled hypertension, serious cardiac arrhythmia requiring medication, or psychiatric illness/social situations that would limit compliance with study requirements.
* Patients with a known sensitivity to any of the products to be administered during treatment.
* Patients unable to undergo MRI of the brain.
* Women who are pregnant or lactating. Women of childbearing potential must have a negative serum or urine pregnancy test performed within 7 days prior to start of treatment. Women of childbearing potential or men with partners of childbearing potential must use effective birth control measures during treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 118 (Actual)
Dates: Start 2017-01-20 (Actual); Primary Completion 2024-12-30 (Actual); Study Completion 2024-12-30 (Actual)

PRIMARY OUTCOMES:
Overall Survival | Every 30 days from randomization until patient death
  Length of time from start of treatment (Day 1) until patient death

SECONDARY OUTCOMES:
Estimate Progression-free Survival | Every 30 days from randomization until disease progression or patient death, whichever occurs earlier
  Time from start of treatment (Day 1) until to the first occurrence of progression or patient death, whichever occurs first
Estimate Median Progression-Free Survival | Every 30 days from randomization until disease progression or patient death, whichever occurs earlier
  The median length of time from start of treatment (Day 1) until to the first occurrence of progression or patient death, whichever occurs first
Estimate Median Overall Survival | Every 30 days from randomization until patient death
  The median length of time from start of treatment (Day 1) until patient death
Estimate Overall Response Rate | Every 42 days from randomization to achievement of either complete response (CR) or partial response (PR)
  Overall number of tumor complete response (CR) or partial response (PR) determined via MRI assessment
Estimate Duration of Response | Every 42 days from the first occurrence of a documented, objective response until the time of relapse or patient death
  Length of time tumor continues to demonstrate either complete response (CR) or partial response (PR) via MRI assessment
Safety evaluation of VAL-083 in patients | From randomization up to 28 days following last study treatment
  To confirm safety and tolerability of VAL-083 using NCI CTCAE v.4 to assess adverse events
Patient Quality of Life Assessment | Every 42 days from randomization until disease progression
  MD Anderson Symptom Inventory-Brain Tumor Module (MDASI-BT)
Plasma Pharmacokinetics | Cycle 1 Day 1 predose, 15 ± 5 min, 30 ± 5 min, 60 ± 10 min, 120 ± 10 min, 240 ± 15 min, and 360 ± 15 min after the end of the of iv infusion of VAL-083
  PK profile and dose-exposure relationship of VAL-083

CONTACTS AND LOCATIONS:
Overall Officials: Barbara O'Brien, M.D., Principal Investigator — University of Texas, MDAnderson Cancer Center, Houston, Texas, USA 77030
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No
The Clinical Study Report for this trial will be prepared and provided to U.S. F.D.A. as required by applicable regulatory requirement(s). Each participating trial investigator will be provided a copy their patient data captured in the electronic data base for this trial.